CLINICAL TRIAL: NCT03185078
Title: Effect of Different Doses of Extracorporeal Shock Wave Therapy on Diabetes Related Frozen Shoulder
Brief Title: Extracorporeal Shock Wave Therapy on Diabetes Related Frozen Shoulder
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Collaborators: Medipol University (Other)
Responsible Party: Principal Investigator, Tülay Çevik, PT, MSc, Okan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Okan University
Record Dates: First submitted 2017-05-29; First posted 2017-06-14 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Frozen Shoulder; Diabetes Mellitus
Keywords: physical therapy; ESWT
MeSH Terms: conditions — Bursitis; Diabetes Mellitus | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active Comparator: Low density ESWT Application (Experimental): ESWT application will be done at energy density of 0.12 mJ/mm2.
  Interventions: Device: Extracorporeal Shock Wave Therapy; Other: Placebo ESWT
- Active Comparator: High density ESWT Application (Experimental): ESWT application will be done at an energy density of 0.3 mJ/mm2.
  Interventions: Device: Extracorporeal Shock Wave Therapy; Other: Placebo ESWT
- Control (Sham Comparator): The ESWT application will be executed when the ESWT application is in the off position. During application, pre-recorded sound beats will be played to the treatment group.
  Interventions: Other: Placebo ESWT

INTERVENTIONS:
Device: Extracorporeal Shock Wave Therapy — Extracorporeal shock wave therapy (ESWT) is a treatment method for the application of single-pulse acoustic pressure waves generated by sudden changes in pressure by creating shock waves with piezoelectric, electrohydraulic and electromagnetic systems. It has been reported that ESWT treatment is effective in the treatment of pain with hyperstimulation analgesia by inhibiting afferent pain receptors, and also improve angiogenesis and restore and reorganize the musculoskeletal system
  Arms: Active Comparator: High density ESWT Application; Active Comparator: Low density ESWT Application
Other: Placebo ESWT — In the placebo application, rESWT device was switched on but without pressing the pedal during the same session period. The applicator was positioned to be the same as the other groups.

SUMMARY:
The aim of this study is to observe the changes in the combined ESWT application and physiotherapy program in the frozen shoulder pathology associated with diabetes. Different treatment approaches will try to identify the most effective treatment method. Changes in muscle tone, pain, range of motion and functionallity will be observed with ESWT treatment. For the first time placebo-controlled research is being conducted with different doses of ESWT in our country and in the World literature. In this way the lower floor of the further work to be done will be established.

DETAILED DESCRIPTION:
The study will be performed with participants who has diabetic frozen shoulder diagnosis after clinical examination and imaging procedures performed, held at Okan University Hospital, Physical Therapy and Rehabilitation Clinic. Data will be recorded with the shoulder evaluation form in the study and cases will be divided into three groups with simple randomization method. The initial range of motion of the participants will be evaluated bilaterally using an electro-goniometer. The muscle tone evaluation will be made with MyotonPro. Muscle strength assessment will be performed with the MicroFET2 dynamometer at the appropriate measurement positions. Participants' pain assessment will be done in the rest, activity and night pain using the Visual Analog Scale. The Shoulder Pain Disability Scale will be used to assess participants' shoulder function. The short-form-36 questionnaire will be used evaluating the quality of life. Physiotherapy application will be applied to all three groups in the form of standard treatment protocol, duration and number. For the first group ESWT application will be done at energy density of 0.12 mJ/mm2, in the second group, at an energy density of 0.3 mJ/mm2, for the third group application will be done as sham ESWT. The ESWT will be administered once a week and in two separate sessions of 2000 strokes. After initial measurements, re-evaluations will be done in the fourth and sixth weeks. The statistics will be analyzed by appropriate methods.

ELIGIBILITY:
Sex: No limit on eligibility based on the sex of participants.

Gender: Eligibility is not based on gender.

Age Limits:

Minimum Age: 30 years Maximum Age: 65

Inclusion Criteria:

Pain in the shoulder joint longer than for six weeks The shoulder joint movements of cases at least two of the abduction, flexion, external rotation, and internal rotation movements with a limitation of motion > 50% Differentiated from other pathologies according to shoulder MRI results

Exclusion Criteria:

Limitation of pain due to cervical radiculopathy Rotator cuff massive tears Recurrent subluxation Trauma or patients with active infection Using cardiac pills, patients Blood coagulation disorders Neurologic causes-restriction of movement in shoulder joint due to cerebrovascular pathologies, Limitation of movement due to rheumatic causes

Sampling Method: Simple random sampling

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
SPADI | Change from baseline shoulder functionality, at the 4th week and at the 6th week.
  The Shoulder Pain and Disability Index. The SPADI contains 13 items that assess two domains; a 5-item subscale that measures pain and an 8-item subscale that measures disability.
VAS | Change will be assessed about pain, at the 4th week and at the 6th week from baseline
  Visual Analog Scale In the study, the chart on the 10 cm length of the diseased pain
  0: painless; 10: It was told that it was unbearable pain.
  Patients were asked to mark the appropriate interval for their pain. The point marked by the patient was measured and recorded with the aid of a ruler

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Okan University Hospital, Istanbul, Tuzla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No